CLINICAL TRIAL: NCT03798639
Title: Randomized, Multi-Institutional Pilot Study of Nivolumab and Radiation Therapy Versus Nivolumab and Ipilimumab as Adjuvant Therapy for Merkel Cell Carcinoma
Brief Title: Nivolumab and Radiation Therapy or Ipilimumab as Adjuvant Therapy in Treating Patients With Merkel Cell Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Claire Verschraegen (Other)
Responsible Party: Sponsor-Investigator, Claire Verschraegen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-18231; NCI-2018-03329 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Merkel Cell Carcinoma; Pathologic Stage IIIA Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIB Merkel Cell Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (nivolumab, radiation therapy) (Experimental): Patients receive nivolumab IV over 30 minutes at week 0. Treatments repeat every 4 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Beginning week 2, patients also receive radiation therapy on Monday-Friday or 5 days per week for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Radiation: Radiation Therapy
- Arm II (nivolumab, ipilimumab) (Active Comparator): Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes at week 0. Treatments repeat every 2 weeks for nivolumab and 6 weeks for ipilimumab for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm II (nivolumab, ipilimumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Radiation: Radiation Therapy — Receive radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
  Arms: Arm I (nivolumab, radiation therapy)

SUMMARY:
This phase I trial studies the side effects and how well nivolumab works when given together with radiation therapy or ipilimumab as adjuvant therapy in treating patients with Merkel cell cancer. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body?s immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays, gamma rays, neutrons, protons or other sources to kill tumor cells and shrink tumors. Giving nivolumab with radiation therapy or ipilimumab after surgery may kill any remaining tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the tolerability of two different experimental immunotherapy regimens in the adjuvant setting in patients with Merkel cell carcinoma (MCC).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability profile of each of the treatment using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

II. To assess the efficacy of each of the treatment arms according to recurrence-free survival (RFS) at one and half years, defined as the time between the date of randomization and the date of first progression (local, regional or distant metastasis) or death (whatever the cause), whichever occurs first.

III. To assess the efficacy of each of the treatment arms according to overall survival (OS) at three years, defined from the time of randomization and the date of death, compared to historical registry control.

EXPLORATORY OBJECTIVES:

I. To explore potential biomarkers, next generation T cell receptor (TCR) sequencing will be performed to identify and longitudinally track individual T cell clones thus granting a comprehensive insight into immunological changes that occur within the tumor and peripheral blood throughout the course of the disease.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive nivolumab intravenously (IV) over 30 minutes at week 0. Treatments repeat every 4 weeks for 1 year in the absence of disease progression or unacceptable toxicity. Beginning week 2, patients also receive radiation therapy on Monday-Friday or 5 days per week for 6 weeks in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes at week 0. Treatments repeat every 2 weeks for nivolumab and 6 weeks for ipilimumab for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to understand and give written informed consent and comply with all study related procedures
* All patients should undergo definitive surgical resection, including when possible sentinel lymph node dissection
* Patients must have recovered after any recent surgery and be ambulatory
* Have node positive disease (stage pIIIA or pIIIB) +/- extracapsular extension
* Have node negative disease and any of the following high risk features

  * Tumor size >= 2 cm
  * Margins =< 1-2 cm and re-resection is not possible
  * Evidence of perineural or lymphovascular invasion
* Human immunodeficiency virus (HIV) patients with undetectable viral load and CD4+ T-cell counts >= 350 cells/uL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count (ANC) >= 1,500/mcL (performed within 16 days of treatment initiation)
* Platelets >= 100,000/mcL in the absence of transfusion support within 7 days of determining eligibility (performed within 16 days of treatment initiation)
* Hemoglobin >= 8 g/dL (performed within 16 days of treatment initiation)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR Measured or calculated creatinine clearance >= 40 mL/min creatinine clearance (performed within 16 days of treatment initiation) (Glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl])

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 x ULN OR Except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 x ULN (performed within 16 days of treatment initiation)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x ULN (performed within 16 days of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy at screening and within 24 hours prior to receiving the first dose of study medication and then every 4 weeks while on treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 5 months after the last dose of study medication. Subjects should agree to ongoing pregnancy testing during the course of the study and after the end of study therapy. Female subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy. Males must refrain from donating sperm during study participation and for 7 months after the last dose of study medication. Female subject should agree to use an adequate method of contraception starting with the first dose of study therapy through 5 months after the last dose of study therapy

Exclusion Criteria:

* Has known distant metastatic MCC
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to any study agents
* Have received prior immunotherapy with any PD-1/PDL-1 inhibitors or CTLA-4 antibodies at any time in the past
* Has had prior chemotherapy or radiation therapy for treatment of MCC
* Has a clinically significant medical condition, which in the judgment of the attending physician would contraindicate immunotherapy or radiotherapy, such as serious autoimmune disease, hypersensitivity to investigational product or any component in its formulations, per Food and Drug Administration (FDA) prescription notice
* Subjects with prior history of non-Merkel cell carcinoma malignancies are excluded except

  * Adequately treated basal cell, squamous cell skin cancer, chronic lymphocytic leukemia (CLL) or other indolent malignancies not requiring therapy (ie. active surveillance)
  * Adequately treated malignancies and patient has been in complete remission for at least two years
  * Patients with history of breast cancer and no evidence of disease on hormonal therapy to prevent recurrence
  * Patients with prostate cancer on adjuvant hormonal therapy with undetectable PSA are eligible
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization will be excluded. Inhaled or topical steroids are permitted in the absence of active autoimmune disease
* Has an active infection requiring intravenous systemic therapy
* Solid organ transplant recipients and patients with concurrent hematological malignancies including thymomas, leukemias (other than CLL) and lymphomas actively undergoing treatment or completed < 5 years prior
* Clinically significant cardiovascular disease with uncontrolled arrhythmia, New York Association class 3 or 4 congestive heart failure, history of myocardial infarction within 6 months, or prolonged corrected QT (QTc) > 500 msec
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients completing 12 months of treatment | Up to 12 months
  Will be estimated along with the 95% confidence interval for each arm based on the binomial distribution.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) one and half years | Time between the date of randomization and the date of first progression (local, regional or distant metastasis) or death (whatever the cause), assessed up to one and half years.
  Kaplan-Meier curves will be generated to summarize the secondary outcomes, RFS and overall survival (OS), for each arm; the differences between groups in terms of hazard ratio for OS/RFS will also be estimated.
Overall survival at three years | Time from randomization to the date of death, assessed up to 3 years
  Kaplan-Meier curves will be generated to summarize the secondary outcomes, RFS and OS, for each arm; the differences between groups in terms of hazard ratio for OS/RFS will also be estimated.
Incidence of adverse events (AEs) | Up to 3 years post treatment
  Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Side effects will be summarized by each treatment group.

OTHER OUTCOMES:
T cell analysis | Baseline up to 3 years post treatment
  TT cell analysis will be performed using peripheral blood at regular time points during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Claire Verschraegen, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu